CLINICAL TRIAL: NCT04483284
Title: Exploratory Clinical Study of TACE Combined With Camrelizumab in the Treatment of BCLC Stage B and Stage C Hepatocellular Carcinoma
Brief Title: Study of TACE Combined With Camrelizumab in the Treatment of HCC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-Ⅱ-003
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined with Camrelizumab (Experimental): Camrelizumab（200mg q3w ivgtt）combined with TACE,the interval between TACE treatment and Carilizumab is not less than 7 days.
  Interventions: Drug: TACE combined with Camrelizumab; Procedure: TACE plus Camrelizumab

INTERVENTIONS:
Drug: TACE combined with Camrelizumab — Camrelizumab(200mg q3w ivgtt) combined with TACE
  Other Names: TACE plus Camrelizumab
Procedure: TACE plus Camrelizumab — Camrelizumab(200mg q3w ivgtt) combined with TACE

SUMMARY:
It is an exploratory clinical study aimed to evaluate the efficacy and safety of TACE combined with Camrelizumab in the treatment of patients with BCLC stage B and C HCC.Treatment will continue until disease progression or intolerable toxicity or patients withdrawal of consent,and the target sample size is 60 individuals.

DETAILED DESCRIPTION:
This is a prospective, single-center and single-arm exploratory clinical study designed to evaluate the efficacy and safety of TACE combined with Camrelizumab in the treatment of patients with BCLC stage B and C hepatocellular carcinoma.Treatment will continue until disease progression or intolerable toxicity or patients withdrawal of consent,and the target sample size is 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients voluntarily entered the study and signed informed consent form (ICF) 2. Age: 18 - 80 years old and life expectancy of at least 12 weeks.; 3. Clinically or histologically diagnosed as HCC; 4. There are measurable lesions that meet the RECIST1.1 standard on the baseline imaging examination; 5. Child-pugh classification A or B (score < 7); 6. The BCLC stage is stage B or C, and it is unable or unwilling to undergo surgical treatment; 7. ECOG : 0 ~ 1 ; 8. No previous immune checkpoint inhibitor treatment (including PD-1 / PD-L1 antibody and CTLA-4 inhibitor); 9. HBV-deoxyribonucleic acid (DNA) must be <500IU / mL, and receive at least 14 days of anti-HBV treatment before the start of study treatment Treatment;

Exclusion Criteria:

* 1. History of treatment with any local treatment (exception of liver transplantation), systemic .anti-cancer therapy, or immunotherapy; 2. Those whose tumor thrombus reaches or exceeds the main portal vein; 3. Existing or concurrently suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma; 4. There is any active autoimmune disease or has a history of autoimmune disease and may relapse; 5. Use strong CYP3A4 / CYP2C19 inducers including rifampicin and Hypericum perforatum or strong CYP3A4 / CYP2C19 inhibitors within 14 days before starting the study treatment; 6. Known history of severe allergy to any monoclonal antibody; 7. Patients who are going to undergo or have undergone organ or allogeneic bone marrow transplantation; 8. Non-compliance with TACE or Camrelizumab; 9. Moderate and severe ascites with clinical symptoms require therapeutic puncture, drainage, or Childa-Pugh score> 2 (except imaging only shows a small amount of ascites but not accompanied by clinical symptoms); uncontrolled or moderate and Above pleural effusion and pericardial effusion; 10. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the start of the study treatment; 11. Thrombosis or embolism occurred within 6 months before the start of study treatment, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction, pulmonary embolism, etc.) 12. Known inherited or acquired bleeding or thrombophilia ; currently or recently (10 days prior to the start of study treatment) have used full dose oral or Injection of anticoagulant drugs or thrombolytic drugs (prophylactic use of low-dose aspirin and low molecular weight heparin); 13. Major vascular disease within 6 months before the study treatment; 22. Past or present central nervous system metastasis; 14. Metastatic diseases involving major airways or blood vessels or a large mediastinal tumor mass in the center (<30 mm from the crest) 15. Those with a history of hepatic encephalopathy; 16. Palliative radiotherapy for non-target lesions allowed for symptom control must be completed at least 2 weeks before the start of study treatment. Adverse events caused by radiotherapy have not recovered to ≤CTCAE level 1; 17. There were severe infections within 4 weeks before starting the study treatment; 18. Patients with congenital or acquired immune deficiency (such as those infected with HIV); 19. Co-infection with hepatitis B and C; 20. For patients with bone metastases, the palliative radiotherapy area> 5% bone marrow area received within 4 weeks before participating in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | an expected average of 8 months
  the time from enrollment to the first disease progression or death from any cause

SECONDARY OUTCOMES:
Time to progression | An expected average of 8 months
  the time from enrollment to the first disease progression
Overall survival | An expected average of 24 months
  the time from enrollment to the death from any cause
Objective response rate | An expected average of 8 months
  evaluated by investigators with mRECIST
Disease control rate | An expected average of 8 months
  evaluated by investigators with mRECIST
Duration of response | An expected average of 8 months
  evaluated by investigators with mRECIST
The incidence of AEs and SAEs by NCI-CTCAE v5.0 | An expected average of 8 months
  Safety index

CONTACTS AND LOCATIONS:
Overall Officials: Yan zhiping, M.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Department of Interventional Radiology, Zhongshan Hospital, Fudan University., Shanghai, Shanghai Municipality, China